CLINICAL TRIAL: NCT03279991
Title: Neuromed- Integrated Health Life Platform and Biobank
Acronym: PLATONE
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Licia Iacoviello, Professor, Neuromed IRCCS
Other Study IDs: 51/17
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases; Neuro-Degenerative Disease; Cancer; Pregnancy
Keywords: biobank; chronic disease; omics; big data; 4 P medicine
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The residual portion of biological withdrawals and materials normally used for the patient's therapeutic diagnostic route ( blood, urine, any fragments of biopsy tissue, surgical finds, umbilical cord, placenta sections, cephalorachidian fluid etc). In order to carry out any genetic-molecular investigations, DNA and DNA from these biological fluids and tissues will be extracted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to create a digital platform for personal, clinical, diagnostic and environmental data collection, management and analysis of patients with cardiovascular and neurological disease or cancer admitted to the Neuromed Group clinics, associated with a biobanks of biological fluids and human tissues and a biotechnological platform for "omics" analysis, to encourage personalized, preventative and predictive care.

DETAILED DESCRIPTION:
There is a need for a change of vision in health care that could become a key innovation point for digital medicine in the future, a sort of Copernican revolution: the starting point is no longer the disease, but the patient around whom pathologies and risk factors rotate, not as distinct and uniquely defined entities, but as communicating and interconnected possibilities that define their form only in relation to the individual, his genome, his personality, his habits of life and the environment in which he lives. From these interactions, a personalized, dynamic, integrated, and continuous diagnostic and therapeutic pathway is created that accompanies the person not only in the stage of the disease but also in the previous and subsequent phases, becoming a way of life oriented towards the health of the person rather than a way to cure a disease.

An Integrated Health Life Platform enables you to develop an interactive healthcare health model among all actors who manage the health of the person, healthcare professionals in the area, and hospitals, caregivers, and community through the integration of remote monitoring of data with A virtual community.

The platform is thought not as a pure aggregation of data, but as a digital hub centered on the patient, with his (clinical and personal) data, but also the environment in which he lives, his behaviors, accessibility to services and The relationships that come to them and from them. The platform aims to effectively integrate self management, personalization of the path, and co-production of health, demonstrating that these three key dimensions of care are mutually reinforcing.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Older than 18 years
* Cardiovascular disease
* neurodegenerative disease
* Cancer
* Pregnancy

Exclusion Criteria:

* Inability to understand and to want
* Refusal to sign the informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in the Neuromed group clinics who will have signed informed consent
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Biological sample bank | baseline
  A repository of biological samples, "Neurobiobank", from patients who will join the project, will be organised at the biotechnology park of Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) Neuromed of Pozzilli under the responsibility of the experienced staff at the Department of Epidemiology and Prevention.
Integrated health-life big data platform | baseline
  Analytical tools will be developped for integrating structured and unstructured patients data sets and derive actionable information from their observed interrelationships.
omics analysis | baseline
  Measure of genomic, epigenetic and proteomic fingerprint of recruited patients
Four P (4P) medicine | Baseline
  Identification of patterns within the health data that correlate with disease or wellness and create personalised pathway of prevention and care.

CONTACTS AND LOCATIONS:
Overall Officials: licia Iacoviello, MD, PhD, Study Chair — IRCCS Neuromed
Locations (1):
- IRCCS INM Neuromed, Department of Epidemiology and Prevention, Pozzilli, IS, Italy

IPD SHARING:
Plan to Share IPD: Yes
submission of a research proposal form to be approved by the Moli-sani scientific committee and signature of a research agreement.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Upon request
Access Criteria: Approval by the Moli-sani study Scientific committee

REFERENCES:
- [Background] GBD 2015 SDG Collaborators. Measuring the health-related Sustainable Development Goals in 188 countries: a baseline analysis from the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1813-1850. doi: 10.1016/S0140-6736(16)31467-2. Epub 2016 Sep 21. PMID 27665228
- [Background] Iacoviello L, De Curtis A, Donati MB, de Gaetano G. Biobanks for cardiovascular epidemiology and prevention. Future Cardiol. 2014 Mar;10(2):243-54. doi: 10.2217/fca.13.110. PMID 24762252
- [Background] Fortier I, Doiron D, Burton P, Raina P. Invited commentary: consolidating data harmonization--how to obtain quality and applicability? Am J Epidemiol. 2011 Aug 1;174(3):261-4; author reply 265-6. doi: 10.1093/aje/kwr194. Epub 2011 Jul 11. PMID 21749975
- [Background] Kim DH, Kim YS, Son NI, Kang CK, Kim AR. Recent omics technologies and their emerging applications for personalised medicine. IET Syst Biol. 2017 Jun;11(3):87-98. doi: 10.1049/iet-syb.2016.0016. PMID 28518059
- [Background] Duffy MJ, O'Donovan N, McDermott E, Crown J. Validated biomarkers: The key to precision treatment in patients with breast cancer. Breast. 2016 Oct;29:192-201. doi: 10.1016/j.breast.2016.07.009. Epub 2016 Aug 9. PMID 27521224